CLINICAL TRIAL: NCT01013974
Title: Phase I Study of GSK573719 -A Randomized, Double Blind, Placebo Controlled, Dose Ascending, Single and Repeat Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Inhaled Dose of GSK573719 From a Novel Dry Powder Device in Healthy Japanese Male Subjects
Brief Title: A Study of GSK573719 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113377
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- GSK573719 250 microgram (μg) arm (Experimental): Each subject will receive the first dose of GSK573719 250 μg on Day 1 followed by once daily dosing for 7 days from Day 4 to Day 10 via a novel dry powder inhaler.
  Interventions: Drug: GSK573719 250 μg
- GSK573719 500 μg arm (Experimental): Each subject will receive the first dose of GSK573719 500 μg on Day 1 followed by once daily dosing for 7 days from Day 4 to Day 10 via a novel dry powder inhaler.
  Interventions: Drug: GSK573719 500 μg
- GSK573719 1000 μg arm (Experimental): Each subject will receive the first dose of GSK573719 1000 μg on Day 1 followed by once daily dosing for 7 days from Day 4 to Day 10 via a novel dry powder inhaler.
  Interventions: Drug: GSK573719 1000 μg
- Placebo (Placebo Comparator): Each subject will receive GSK573719 matching placebo on Day 1 followed by once daily dosing for 7 days from Day 4 to Day 10 via a novel dry powder inhaler.
  Interventions: Drug: GSK573719 matching Placebo

INTERVENTIONS:
Drug: GSK573719 250 μg — Strip 1 of the dry powder inhaler will contain GSK573719 250 μg micronized drug with lactose along with magnesium stearate. Strip 2 will contain lactose powder along with magnesium stearate. It will be available as dry off white powder for inhalation.
  Arms: GSK573719 250 microgram (μg) arm
Drug: GSK573719 500 μg — Strip 1 of the dry powder inhaler will contain GSK573719 500 μg micronized drug with lactose along with magnesium stearate. Strip 2 will contain lactose powder along with magnesium stearate. It will be available as dry off white powder for inhalation.
  Arms: GSK573719 500 μg arm
Drug: GSK573719 1000 μg — Strips 1 and 2 of the dry powder inhaler will contain 500 μg each of GSK573719 micronized drug with lactose along with magnesium stearate. It will be available as dry off white powder for inhalation.
  Arms: GSK573719 1000 μg arm
Drug: GSK573719 matching Placebo — Strip 1 and 2 of the dry powder inhaler will contain lactose powder along with magnesium stearate. It will be available as dry off white powder for inhalation.
  Arms: Placebo

SUMMARY:
This is a single centre, randomized, double blind, placebo controlled, single and repeat dose study to investigate the safety, tolerability, and pharmacokinetics of inhaled dose of GSK573719 with lactose and containing magnesium stearate by a novel dry powder device in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy male subjects aged between 20 and 64 years of age inclusive. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies, and other tests.
2. Body weight ≥ 50kg and BMI within the range 18.5-25.0kg/m2 inclusive.
3. Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
4. Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
5. Clinical laboratory tests data obtained at screening meet the following:

   AST(GOT), ALT(GPT), total-bilirubin: below the upper limit of the normal ranges
6. Normal 12-lead EGC finding at screening; QTc(B) interval <450msec
7. A mean blood pressure lower than 140/90mmHg at screening.
8. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
9. Capable of using the novel dry powder inhaler.

Exclusion Criteria:

1. The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
2. The subject is positive for syphilis, HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody.
3. The subject is positive for urine drug screening.
4. The subject has an allergy for any drug or idiosyncrasy
5. The subject has a history of breathing problems (i.e. history of asthmatic symptomatology).
6. The subject has a history of cardiovascular disease.
7. The subject has a significant clinical history or current conditions of glaucoma.
8. The subject has a significant clinical history or current conditions of prostatic hypertrophy.
9. The subject has a history of drug abuse or alcoholism.
10. The subject has a history of cholecystectomy or biliary tract disease.
11. History of regular alcohol consumption exceeding on average, 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 350 mL of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 month of screening.
12. Use of prescription or non-prescription drugs, including CYP3A/PGP inhibitor, vitamins, herbal and dietary supplements (including St John'sWort) within 14 days prior to the first dose of study medication.
13. The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
14. The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months.
15. The subject has an allergy for any drug hypersensitivity to milk protein or the excipients lactose monohydrate and magnesium stearate.
16. The subject has donated a unit of blood ">400 mL" within the previous 4 months or ">200 mL" within the previous 1 month.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10-05 (Actual); Primary Completion 2009-12-18 (Actual); Study Completion 2009-12-18 (Actual)

PRIMARY OUTCOMES:
PK: Cmax, tmax and AUC(0-t)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kagoshima, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113377 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113377?search=study&search_terms=113377#rs
- Available data/document: Dataset Specification: 113377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register